CLINICAL TRIAL: NCT04131842
Title: External Versus Internal Feedback on Biomechanics and Self-reported Function in Patients With Chronic Ankle Instability
Brief Title: External Versus Internal Feedback in Patients With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Charlotte (Other)
Responsible Party: Principal Investigator, Luke Donovan, Assistant Professor, University of North Carolina, Charlotte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRBIS-19-0263
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Ankle Injuries; Ankle Inversion Sprain
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ExFOCUS Visual (Experimental): Participants will complete 12 sessions over 4-weeks of impairment-based rehabilitation that incorporates ankle range of motion, ankle strength, balance, and functional activity exercises. For the balance and functional activity exercises, participants will use traditional instability tools and will receive external focus of attention visual feedback.
  Interventions: Other: External focus of attention visual feedback
- ExFOCUS Auditory (Experimental): Participants will complete 12 sessions over 4-weeks of impairment-based rehabilitation that incorporates ankle range of motion, ankle strength, balance, and functional activity exercises. For the balance and functional activity exercises, participants will use traditional instability tools and will receive auditory feedback.
  Interventions: Other: External focus of attention auditory feedback
- InFOCUS Visual (Experimental): Participants will complete 12 sessions over 4-weeks of impairment-based rehabilitation that incorporates ankle range of motion, ankle strength, balance, and functional activity exercises. For the balance and functional activity exercises, participants will use traditional instability tools and will receive internal focus of attention visual feedback via video.
  Interventions: Other: Internal focus of attention video feedback
- NoFeedback (Active Comparator): Participants will complete 12 sessions over 4-weeks of impairment-based rehabilitation that incorporates ankle range of motion, ankle strength, balance, and functional activity exercises. For the balance and functional activity exercises, participants will use traditional instability tools and receive no feedback.
  Interventions: Other: No feedback

INTERVENTIONS:
Other: External focus of attention visual feedback — Patients will receive external focus of attention visual feedback during the impairment-based rehabilitation program.
  Arms: ExFOCUS Visual
Other: External focus of attention auditory feedback — Patients will receive external focus of attention auditory feedback during the impairment-based rehabilitation program.
  Arms: ExFOCUS Auditory
Other: Internal focus of attention video feedback — Patients will receive internal focus of attention visual feedback during the impairment-based rehabilitation program.
  Arms: InFOCUS Visual
Other: No feedback — Patients will receive no feedback during the impairment-based rehabilitation program.
  Arms: NoFeedback

SUMMARY:
Although altered biomechanics has been well documented as an impairment associated with chronic ankle instability (CAI), effective interventions targeting biomechanics with long-term outcomes measuring patient-reported outcomes (PROs) are absent. Evidence suggests that external focus of attention (ExFOCUS), internal focus of attention (InFOCUS) feedback, and auditory feedback during movement training can alter biomechanics in other patient populations, with ExFOCUS and auditory enhancing retention of learned biomechanics. Therefore, this randomized controlled trial will determine if a 4-week (12 session) impairment-based rehabilitation program that includes feedback (ExFOCUS or InFOCUS or Auditory) can (1) decrease ankle inversion kinematics and lateral plantar pressure during walking and (2) improve self-reported function.

ELIGIBILITY:
Inclusion Criteria:

* Characterized as having chronic ankle instability (CAI) by reporting a history of recurrent ankle sprains, with the first sprain occurring longer than 12 months ago. Participants will have lingering symptoms, and disability, but have not actively sought treatment for their CAI.
* All participants will be physically active: Participating in some form of physical activity for at least 20 min per day, three times per week.

Exclusion Criteria:

* Neurological or vestibular disorders affecting balance
* Currently seeking medical care for CAI
* History of ankle surgery
* History of ankle sprain within the past 6 weeks
* History of other musculoskeletal injuries within the past 6 weeks
* Current/previous self-reported disability due to lower extremity pathology that may adversely affect neuromuscular function

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in lower extremity kinematics and kinetics during walking | Immediate post-intervention, 1-month post-intervention, 3-months post-intervention
  Ankle, knee, and hip motion and moments during walking measured by a 3D motion capture system and in shoe plantar pressure system
Changes from baseline in self-reported ankle function | Immediate post-intervention, 1-month post-intervention, 3-months post-intervention
  Changes from baseline in self-reported function as measured by the Foot and Ankle Ability Measure (FAAM) Activities of Daily Living and Sport questionnaire. Scores range from 100% (no decrease in function) to 0% (complete loss of function).

SECONDARY OUTCOMES:
Changes from baseline in ankle range of motion measured in degrees | Immediate post-intervention, 1-month post-intervention, 3-months post-intervention
  Four different ankle ranges of motion will be measured
Changes from baseline in ankle maximum voluntary isometric strength | Immediate post-intervention, 1-month post-intervention, 3-months post-intervention
  Ankle maximum voluntary isometric strength will be measured during four different ankle positions using a hand-held dynamometer.
Changes from baseline in static and dynamic balance | Immediate post-intervention, 1-month post-intervention, 3-months post-intervention
  Static balance will be measured via a force plate and dynamic balance will be measured using the Star Excursion Balance Test

CONTACTS AND LOCATIONS:
Locations (1):
- UNC Charlotte, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No